CLINICAL TRIAL: NCT03263559
Title: Reduced Intensity Conditioning for Haploidentical Bone Marrow Transplantation in Patients With Symptomatic Sickle Cell Disease. (BMTCTN1507)
Brief Title: Haploidentical Bone Marrow Transplantation in Sickle Cell Patients (BMTCTN1507)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN1507; 2U10HL069294-11 (NIH); 5U24CA076518 (NIH)
Record Dates: First submitted 2017-08-24; First posted 2017-08-28 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Sickle Cell Disease
Keywords: Reduced Intensity Conditioning; Haploidentical; Bone Marrow; Transplant; Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea; Antilymphocyte Serum; thymoglobulin; Thiotepa; Drug Therapy; fludarabine; fludarabine phosphate; Cyclophosphamide; Whole-Body Irradiation; Mesna

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Haploidentical Transplantation (Experimental): A conditioning regimen with Hydroxyurea, rabbit-ATG, Thiotepa, Fludarabine, Cyclophosphamide, Total Body Irradiation, and Mesna will be administered prior to Haploidentical Bone Marrow Transplantation.
  Interventions: Procedure: Haploidentical Bone Marrow Transplantation; Drug: Hydroxyurea; Drug: Rabbit-ATG; Drug: Thiotepa; Drug: Fludarabine; Drug: Cyclophosphamide; Radiation: Total Body Irradiation; Drug: Mesna

INTERVENTIONS:
Procedure: Haploidentical Bone Marrow Transplantation — Eligible patients with a first degree Human Leukocyte Antigen (HLA)- haploidentical donor will undergo Haploidentical bone marrow transplantation at Day 0 with non T-cell depleted bone marrow. For Graft-vs-Host Disease (GVHD) prophylaxis, patients will be given sirolimus and mycophenolate mofetil beginning on Day +5.
Drug: Hydroxyurea — HU will be given daily at 30mg/kg from Day -70 through Day -10.
  Other Names: Hydrea; Droxia
Drug: Rabbit-ATG — Rabbit-ATG (rATG) will be given at 0.5mg/kg on Day -9, and at 2.0mg/kg on Day -8 and Day -7.
  Other Names: Thymoglobulin
Drug: Thiotepa — Thiotepa will be given at 10mg/kg on Day -7
  Other Names: Chemo
Drug: Fludarabine — Fludarabine will be given at 30mg/m2 from Day -6 to Day -2
  Other Names: Fludara
Drug: Cyclophosphamide — Cyclophosphamide will be given at 14.5mg/kg on Day -6 and Day -5, and at 50 mg/kg on Days +3 and +4.
  Other Names: Cytoxan®
Radiation: Total Body Irradiation — Total Body Irradiation will be given at 200cGy on Day -1
  Other Names: TBI
Drug: Mesna — Mesna will be given at 40mg/kg on Days +3 and +4
  Other Names: Mesnex

SUMMARY:
This is a Phase II, single arm, multi-center trial, designed to estimate the efficacy and toxicity of haploidentical bone marrow transplantation (BMT) in patients with sickle cell disease (SCD). Based on their age and entry criteria patients are stratified into two groups: (1) children with severe SCD; and (2) adults with severe SCD.

DETAILED DESCRIPTION:
This study is designed as a Phase II multi-center trial to determine the feasibility of achieving a high rate of event-free survival (EFS) at 2 years post transplant using pre-conditioning hydroxyurea (HU) with a conditioning regimen that consists of a combination of Thymoglobulin/Cyclophosphamide/Fludarabine/Thiotepa with post-grafting high-dose cyclophosphamide in patients with severe SCD who have HLA-haploidentical donors. EFS is defined as survival without a qualifying event. This is a single arm study in which participants will be enrolled into one of two strata. The first stratum will be restricted to children who have stroke and 40 children will be enrolled in this stratum. The second stratum will consist of adult patients with severe sickle cell disease and 40 participants will be enrolled in this stratum.

ELIGIBILITY:
Inclusion Criteria:

Adequate physical function as measured by all of the following:

1. A Karnofsky/Lansky performance score of ≥ 60.
2. Cardiac function: Left ventricular ejection fraction (LVEF) > 40%; or LV shortening fraction > 26% by cardiac echocardiogram or by Multi Gated Acquisition Scan (MUGA) scan.
3. Pulmonary function: Pulse oximetry with a baseline O2 saturation of ≥ 85% and Diffusing capacity of the lung for carbon monoxide (DLCO) > 40% (corrected for hemoglobin).
4. Renal function: Serum creatinine ≤ 1.5 x upper limit of normal for age and estimated or measured creatinine clearance ≥ 70 mL/min/1.73 m²
5. Hepatic function:

   1. Serum conjugated (direct) bilirubin < 2x upper limit of normal for age as per local laboratory. Participants with hyperbilirubinemia as the result of hyperhemolysis, or a severe drop in hemoglobin post blood transfusion, are not excluded.
   2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 5x upper limit of normal as per local laboratory.
6. Liver MRI using a validated methodology per institutional preference (T2* or R2* or by ferriscan [R2 MRI]) for estimation of hepatic iron content is required for participants who are currently receiving ≥8 packed red blood cell transfusions per year for ≥1 year or have received ≥20 packed red blood cell transfusions (lifetime cumulative). Participants who have hepatic iron content ≥ 10 mg Fe/g liver dry weight by liver MRI must have a Gastroenterology/hepatology consultation with liver biopsy and histological examination including documentation of the absence of cirrhosis, bridging fibrosis, and active hepatitis.
7. Participants must be HLA typed at high resolution using DNA based typing at HLA-A, -B, -C, DRB1, and have available:

   An HLA haploidentical first degree relative donor (parents, siblings or half siblings, or children) with 2, 3, or 4 (out of 8) HLA-mismatches who is willing and able to donate bone marrow. A unidirectional mismatch in either the graft versus host or host versus graft direction is considered a mismatch. The donor and recipient must be HLA identical for at least one antigen (using high resolution DNA based typing) at the following genetic loci: HLA-A, HLA-B, HLA-C, and HLA-DRB1. Fulfillment of this criterion shall be considered sufficient evidence that the donor and recipient share one HLA haplotype, and typing of additional family members is not required. Confirmatory donor HLA typing must be completed < 100 days prior to Segment A enrollment
8. Umbilical cord blood or peripheral blood stem cell donors will not be accepted.

Inclusion Criteria for Stratum 1: Children Ages 5.00 - 14.99 years of age at enrollment

1. Age 5.00 - 14.99 years at Segment A enrollment
2. Participants with sickle cell anemiam disease (Hb SS or Sß° Thalassemia) who have one or more of the following:

   1. A neurological event resulting in focal neurologic deficits that lasted ≥ 24 hours (classical clinical definition of stroke, not requiring imaging studies of the brain) OR a focal neurological event resulting in abnormalities on T2-weighted or FLAIR images using a MRI scan, indicative of an acute infarct, with no other reasonable medical explanation (definition of a stroke supported with MRI imaging scans of the brain), OR both.
   2. Abnormal transcranial Doppler (TCD) measurement with a timed average maximum mean velocity of at least 200 cm/sec in the terminal portion of the internal carotid or proximal portion of middle cerebral artery or if the imaging TCD method is used > 185 cm/sec plus evidence of intracranial vasculopathy.
   3. Silent Cerebral Infarct defined as an infarct-like lesion based on an MRI signal abnormality at least 3 mm in one dimension and visible in two planes on FLAIR or T2-weighted images (or similar image with 3D imaging) and documented neurological examination performed by a neurologist demonstrating the participant has a normal neurologic examination or an abnormality on examination that could not be explained by the location of the brain lesion(s).
   4. Acute severe vaso-occlusive pain episodes requiring hospitalization and recalcitrant to maximum medical therapy. Episodes of pain to be adjudicated by selected committee.
   5. One acute chest syndrome episode resulting in intensive care admission requiring non-mechanical ventilatory support: simple nasal cannula, face mask that requires oxygen content (venti mask, non-rebreather), simple nasal cannula, face mask O2(e.g. ventimask, rebreather), CPAP, SiPAP, BiPAP, high flow nasal cannula (HFNC) or invasive mechanical ventilatory support (delivered by ETT or trach).
   6. Right heart catheterization confirmed pulmonary artery pressure >25 mmHG or mean pulmonary vascular resistance 206(57-421) dyn·s·cm-5
   7. Essential hypertension on antihypertensive medications >95% upper limit of normal age (as defined according to the American Academy of Pediatrics)
   8. Recurrent priapism (episodes lasting at least 4 hours at least twice in the last 12 months or 3 times in the last 24 months) recalcitrant to medical treatment or unable to use hydroxyurea due to SCD phenotype with the approval of the adjudication committee

Inclusion Criteria for Stratum 2: Adults Ages 15.00 - 45.99 at enrollment

Participants with sickle cell anemia (Hb SS or Sß° Thalassemia) who are 15.00 - 45.99 years of age at enrollment AND who have one or more of the following:

1. Age 15.00 - 45.99 years at Segment A enrollment
2. Participants with sickle cell anemia (Hb SS or Sß° Thalassemia) who have one or more of the following:

   1. A neurological event resulting in focal neurologic deficits that lasted ≥ 24 hours (classical clinical definition of stroke, not requiring imaging studies of the brain) OR a focal neurological event resulting in abnormalities on T2-weighted or FLAIR images using a MRI scan, indicative of an acute infarct, with no other reasonable medical explanation (definition of a stroke supported with MRI imaging scans of the brain), OR both.
   2. History of two or more episodes of acute chest syndrome (ACS) in the 2-year period preceding enrollment despite the institution of supportive care measures (i.e. asthma therapy and/or hydroxyurea);
   3. History of three or more severe vaso-occlusive pain crises per year in the 2-year period preceding enrollment despite the institution of supportive care measures (i.e. a pain management plan and/or treatment with hydroxyurea); painful episodes related to priapism, osteonecrosis or any sickle-related complication are acceptable;
   4. Administration of regular RBC transfusion therapy, defined as receiving ≥8 packed red blood cell transfusions per year for ≥1 year in the 12 months before enrollment to prevent vaso-occlusive clinical complications (i.e. pain, stroke, and acute chest syndrome);
   5. An echocardiographic finding of tricuspid valve regurgitant jet velocity (TRJV) ≥ 2.7 m/sec.

Exclusion Criteria:

1. Participants who have an HLA-matched sibling who is able and willing to donate bone marrow. Patients with a HLA-matched unrelated donor are not excluded.
2. Uncontrolled bacterial, viral or fungal infection in the 6 weeks before enrollment (currently taking medication with evidence of progression of clinical symptoms or radiologic findings).
3. Evidence of HIV infection or known HIV positive serology.
4. Participants who have received a previous hematopoetic cell transplant (HCT).
5. Participants who have had an Encephaloduroarteriosynangiosis (EDAS) procedure in the 6 months prior to enrollment
6. Participants who have received a prior solid organ transplant
7. Participants who have participated in another clinical trial in which the patient received an investigational or off-label use of a drug or device within 3 months of enrollment.
8. Females who are pregnant or breastfeeding.
9. Participants with clinically significant, uncontrolled autoimmune disease, requiring active medical management (immunosuppressive therapy or chemotherapy), which, in the judgment of the local Principal Investigator, indicates that the patient could not tolerate transplantation.
10. Females of child bearing potential (to include all female participants > 10 years of age, unless postmenopausal for a minimum of 1 year before the time of consent or surgically sterilized), who do not agree to practice two (2) effective methods of contraception at the same time, or do not agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject, from the time of signing of informed consent through 12 months post-transplant.
11. Males (even if surgical sterilized) who do not agree to practice effective barrier contraception, or who do not agree to practice true abstinence from the time of signing informed consent through 12 months post-transplant.
12. Presence of anti-donor specific HLA antibodies. HLA antibody presence and specificity will be determined by solid phase immunoassays. An anti-donor specific HLA antibody will be considered positive when the mean fluorescence intensity (MFI) is higher than the cut-off defined by each institution. Recommended cut-off values are MFI >1000 for donor specific antibody to HLA-A, -B, and DRB1 and MFI >2000 for HLA-C, DQB1 and DPB1. This must be measured before the final donor selection, and < 100 days before enrollment in Segment A (preferably < 30 days before Segment A enrollment). If MFI >1000 for donor specific antibody to HLA-A, -B, DRB1 and/or MFI >2000 for HLA-C, DQB1 and DPB1, documentation must be submitted to the DCC coordinator for review and approval by a Protocol Chair and/or Protocol Officer prior to enrollment

Ages: 5 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 95 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
Two-Year Post-Transplant Event Free Survival (EFS) | 2 years
  EFS is defined as survival without a qualifying event. Primary graft rejection, secondary graft rejection, second infusion of hematopoietic cells or death will count as events for this endpoint.

SECONDARY OUTCOMES:
Overall Survival | 1 and 2 years
  Death from any cause will be the event and patients will be censored at the date of last contact or two years post-transplant whichever comes first.
One-Year Post-Transplant EFS | 1 year
  EFS is defined as survival without a qualifying event, Primary graft rejection, secondary graft rejection, second infusion of hematopoietic cells or death will count as events for this endpoint.
Graft Rejection | Day 42
  Graft rejection is defined as not having engraftment on or before Day 42 post-transplant. Engraftment is defined as having greater than or equal to 5% donor cells post-transplant, from any molecular chimerism assessment (e.g., unsorted, myeloid, or T-cell) on a peripheral blood or bone marrow aspirate sample.
Chimerism | Days 28, 100, and 180 and at 1 and 2 years
  Characterize donor hematopoietic chimerism in peripheral blood will be assessed.
Disease Recurrence | 2 years
  Disease recurrence is defined as the return of sickle erythropoiesis (in the absence of red blood count transfusion, Hb S level > 70%), or primary or secondary graft rejection, as defined above, or second infusion of hematopoietic cells.
Patient Reported Quality of Life (QoL) | 1 and 2 years
  Health-Related QoL will be measured using patient reported surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, Study Director — Center for International Blood and Marrow Transplant Research
Locations (32):
- United States (32):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - University of Colorado - Denver/Children's Hospital of Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida College of Medicine, Gainesville, Florida
  - Nicklaus Children's Hospital/University of Miami Children's Hospital, Miami, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Northside Hospital, Atlanta, Georgia
  - Riley Children's Hospital at IU Health, Indianapolis, Indiana
  - Indiana University Medical Center, Indianapolis, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Children's Hospital of Michigan, Detroit, Michigan
  - Helen Devos Children's at Spectrum Health, Grand Rapids, Michigan
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University, St. Louis, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Cancer Center, Buffalo, New York
  - Northwell Health/Monter Cancer Center, Lake Success, New York
  - Levine Children's Hospital, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals of Cleveland/Case Western, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Methodist Healthcare/West Cancer Center, Memphis, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Children's Hospital (Baylor), Houston, Texas
  - University of Texas/MD Anderson Cancer Center, Houston, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - The Medical College of Wisconsin, Wauwatosa, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a manuscript and supporting information submitted to NIH BioLINCC (including data dictionaries, case report forms, data submission documentation, documentation for outcomes dataset, etc where indicated).
Supporting Information: Study Protocol, ICF
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Result] Hong S, Horwitz ME. Cures for Sickle Cell Abound - How about Access? NEJM Evid. 2025 Mar;4(3):EVIDe2400428. doi: 10.1056/EVIDe2400428. Epub 2025 Feb 25. No abstract available. PMID 39998301
- [Derived] Kassim AA, Walters MC, Eapen M, Smith M, Logan BR, Solh M, McKinney C, Nieder M, Ross M, Kent M, Abusin GA, Mallhi K, Silva JG, Shaughnessy P, Kanter J, Haines H, Farah R, Khaled YA, Ritzau N, Mendizabal A, Abraham A, Bollard C, Cooke K, de la Fuente J, Hanna R, Horowitz MM, Jordan LC, Bakshi N, Krishnamurti L, Leifer E, Mahadeo KM, Shenoy S, Jones RJ, DeBaun MR, Brodsky RA. Haploidentical Bone Marrow Transplantation for Sickle Cell Disease. NEJM Evid. 2025 Mar;4(3):EVIDoa2400192. doi: 10.1056/EVIDoa2400192. Epub 2025 Feb 25. PMID 39998298
- [Derived] Leonard A, Furstenau D, Abraham A, Darbari DS, Nickel RS, Limerick E, Fitzhugh C, Hsieh M, Tisdale JF. Reduction in vaso-occlusive events following stem cell transplantation in patients with sickle cell disease. Blood Adv. 2023 Jan 24;7(2):227-234. doi: 10.1182/bloodadvances.2022008137. PMID 36240296
- See also: Blood and Marrow Transplant Clinical Trials Network Website — https://bmtctn.net//

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-05-19): https://cdn.clinicaltrials.gov/large-docs/59/NCT03263559/Prot_SAP_ICF_000.pdf